CLINICAL TRIAL: NCT01678170
Title: Clinical Application of Breast Blood-oxygen Functional Imaging Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIH-LPF-201205001
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-05

CONDITIONS: Breast Diseases
Keywords: blood-oxygen functional imaging technology; diagnosis
MeSH Terms: conditions — Breast Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This trial is going to evaluate the value of blood-oxygen functional imaging technology in the diagnosis of breast diseases.

ELIGIBILITY:
Inclusion Criteria:

* female older than 18 years breast lump received breast ultrasound and mammography

Exclusion Criteria:

* After core-needle biopsy or resection After neoadjuvant chemotherapy, radiotherapy or endocrine therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female with breast lump, received breast ultrasound and mammography
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peifang Liu, M.D., Principal Investigator — Department of Breast Imaging, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Breast Imaging, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China